CLINICAL TRIAL: NCT01567696
Title: Defining the Inflammatory Cytokines in Patients With Adverse Reactions to Metal-on-Metal Hip Replacements
Brief Title: Clinical, Radiographic and Laboratory Analysis of Failures of Joint Replacements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Scott Ball, MD, Assistant Clinical Professor; Chief, Joint Reconstruction, University of California, San Diego
Other Study IDs: IIS-000135/11007
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Joint
Keywords: Revision,

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to more fully understand the reason(s) that joint replacement implants fail and to better identify diagnosis and outcome methods both pre-operatively and post-operatively with revision surgery. Analysis of joint replacement failure will include a through analysis of laboratory, radiographic, implant, surgical and demographic data.

DETAILED DESCRIPTION:
To examine all clinical data in patients with failed total hip and total knee replacements including patient demographics (age, sex, comorbidities, etc.), patient clinical data (history and physical exam and lab findings) and including implant specifications and radiographic findings (for implant type, implant size, implant bearing surface type, position, stability, etc.).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* failed hip or knee replacement
* willing to sign informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age, that present with a failed joint replacement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Ball, MD, Principal Investigator — UCSD
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States